CLINICAL TRIAL: NCT04806269
Title: Clinical Application of Continuous Monitoring Data for the Pulse Rate, Exercise, and Symptom Survey by Wearable Device in the Patients With Thyroid Dysfunction
Brief Title: Biosignals by Wearables in Thyroid Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae Hoon Moon, SeoulNUBH, Seoul National University Bundang Hospital
Other Study IDs: B-2012-654-303
Record Dates: First submitted 2021-01-26; First posted 2021-03-19 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Thyrotoxicosis; Hypothyroidism
Keywords: Wearable device; Biosignals; Thyrotoxicosis; Hypothyroidism; Mobile app
MeSH Terms: conditions — Thyrotoxicosis; Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thyroid dysfunction group: Subjects with thyroid dysfunction including thyrotoxicosis and hypothyroidism Subjects who were newly diagnosed or undergoing treatment for thyroid dysfunction can be included in the study.
  Subjects should use a wearable device (Fitbit Inspire 2 TM) and a mobile app (Glandy TM) during the study period.
  Interventions: Device: Fitbit and Glandy
- Control group: Subjects without thyroid dysfunction including thyrotoxicosis and hypothyroidism.
  Subjects should use a wearable device (Fitbit Inspire 2 TM) and a mobile app (Glandy TM) during the study period.
  Interventions: Device: Fitbit and Glandy

INTERVENTIONS:
Device: Fitbit and Glandy — Data collection from wearable devices (Fitbit Inspire 2 TM) and a mobile app (Glandy TM) Fitbit collects user's heart rate, activity, and sleep data. Glandy collects user's subjective symptom scores.

SUMMARY:
This study is a single center observational study to investigate the association between biosignals from wearables and thyroid dysfunction.

DETAILED DESCRIPTION:
An algorithm to predict thyroid dysfunction using heart rate and activity data from wearables was generated based on our previous clinical studies. This study was conducted to collect more data to advance the algorithm.

Patients with thyroid dysfunction including hypothyroidism and thyrotoxicosis were eligible for this study. During the study period, each subject wears a smart band (Fitbit Inspire 2 TM) and gets 3 times of thyroid function tests with 1-month interval. Study participants will use a mobile app (Glandy TM) to collect the symptom scores.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were newly diagnosed as thyroid dysfunction (thyrotoxicosis or hypothyroidism) or undergoing treatment
* Subjects who are able to use wearable devices, smart phones, and mobile apps

Exclusion Criteria:

* Subjects with restrictions on normal activities due to diseases other than thyroid dysfunction
* Subjects who are taking medications affecting heart rate
* Subjects with diseases affecting heart rate (i.e. arrhythmia)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Korean adults (age 18-60) who newly diagnosed as thyroid dysfunction (thyrotoxicosis or hypothyroidism) or undergoing treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
free T4 | visit 2: 1-2 weeks after enrollement (visit 1)
  serum concentration of free T4
free T4 | visit 3 : 4 weeks after visit 2
  serum concentration of free T4
free T4 | visit 4 : 4 weeks after visit 3
  serum concentration of free T4
TSH | visit 2: 1-2 weeks after enrollement (visit 1)
  serum concentration of TSH
TSH | visit 3 : 4 weeks after visit 2
  serum concentration of TSH
TSH | visit 4 : 4 weeks after visit 3
  serum concentration of TSH
heart rate | throughout the study period (average 3 months)
  continuously monitored heart rate by wearable device
Activity_steps (count/min) | throughout the study period (average 3 months)
  continuously monitored steps per minute by wearable device
Sleep_sleep start time (yyyy:mm:dd:hh:mm:ss) | throughout the study period (average 3 months)
  sleep start time extracted from continuously monitored sleep data by wearable device (e.q. 2021:03:15:23:00:00)
Sleep_sleep end time (yyyy:mm:dd:hh:mm:ss) | throughout the study period (average 3 months)
  sleep end time extracted from continuously monitored sleep data by wearable device (e.q. 2021:03:16:06:00:00)
Hyperthyroid symptom scale | visit 2: 1-2 weeks after enrollement (visit 1)
  HSS gives scores from 0 to 40, where higher scores indicate more severe disease. It consists of a 10-item scale that rates nervousness, diaphoresis, heat intolerance, motor activity, tremor, weakness, hyperdynamic precordium, diarrhea, weight loss/appetite, and overall function.
Zulewski's clinical score | visit 2: 1-2 weeks after enrollement (visit 1)
  Clinical scoring system for assessing hypothyroid symptoms and signs (0-12, higher scores indicate more severe)
Hyperthyroid symptom scale | visit 3 : 4 weeks after visit 2
  HSS gives scores from 0 to 40, where higher scores indicate more severe disease. It consists of a 10-item scale that rates nervousness, diaphoresis, heat intolerance, motor activity, tremor, weakness, hyperdynamic precordium, diarrhea, weight loss/appetite, and overall function.
Zulewski's clinical score | visit 3 : 4 weeks after visit 2
  Clinical scoring system for assessing hypothyroid symptoms and signs (0-12, higher scores indicate more severe)
Hyperthyroid symptom scale | visit 4 : 4 weeks after visit 3
  HSS gives scores from 0 to 40, where higher scores indicate more severe disease. It consists of a 10-item scale that rates nervousness, diaphoresis, heat intolerance, motor activity, tremor, weakness, hyperdynamic precordium, diarrhea, weight loss/appetite, and overall function.
Zulewski's clinical score | visit 4 : 4 weeks after visit 3
  Clinical scoring system for assessing hypothyroid symptoms and signs (0-12, higher scores indicate more severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea